CLINICAL TRIAL: NCT03192475
Title: Dissemination of a Diabetes Prevention Program Among Medicare Eligible Older Adults
Brief Title: The Pitt Retiree Study: A Diabetes Prevention Program for Medicare Eligible Older Adults
Acronym: PRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Elizabeth Venditti, Assistant Professor of Psychiatry and Epidemiology, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO12050022
Record Dates: First submitted 2017-06-15; First posted 2017-06-20 (Actual); Results first posted 2019-11-13 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Obesity; Cardiovascular Risk Factor; Eating Behavior; Diet Modification; Physical Activity; Quality of Life; Mobility Limitation
MeSH Terms: conditions — Obesity; Feeding Behavior; Motor Activity; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: An initial (non-randomized) translational Group Lifestyle Balance (GLB) in person, lifestyle intervention designed to mitigate cardiometabolic risk in older adults is delivered to all participants between 0 and 4-months. Subsequently, one-half of the enrolled sample is randomized to either (1) 8-group telephone contacts (8-TC) for the remainder of 12-months; the other one-half is randomized to a newsletter control condition (NC) during this time period.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Lifestyle Balance plus phone contacts (Active Comparator): Group Lifestyle Balance is the core behavioral lifestyle intervention delivered from 0-4 months using an in-person group format. The active comparator receives 8 additional sessions of group interactive telephone contact delivered from 5-12 months
  Interventions: Behavioral: GLB plus phone contacts
- Group Lifestyle Balance plus newsletter contacts (Placebo Comparator): Group Lifestyle Balance is the core behavioral lifestyle intervention delivered from 0-4 months using in-person group format. The placebo comparator receives 4 additional educational newsletters delivered from 5-12 months.
  Interventions: Behavioral: GLB plus newsletter contacts

INTERVENTIONS:
Behavioral: GLB plus phone contacts — GLB is a comprehensive evidence-based lifestyle intervention derived from the Diabetes Prevention Program intensive lifestyle intervention; combines behavior modification strategies and making health changes to diet, physical activity and weight. The active treatment group also receives 8 additional group phone conference calls for social support and problem solving.
  Arms: Group Lifestyle Balance plus phone contacts
Behavioral: GLB plus newsletter contacts — GLB is a comprehensive evidence-based lifestyle intervention derived from the Diabetes Prevention Program intensive lifestyle intervention; combines behavior modification strategies and making health changes to diet, physical activity and weight. The placebo comparator includes 4 additional newsletters only.
  Arms: Group Lifestyle Balance plus newsletter contacts

SUMMARY:
The Pitt Retiree Study (PRS) disseminates a novel, yet practical, diabetes prevention program among Medicare eligible adults in Western Pennsylvania. This study will provide 4, and 12 month outcome data (with a no treatment follow-up assessment at 24 months) to help determine whether a continued contact group telephone intervention is feasible and effective in enhancing health outcomes and physical functional ability in high risk adults (aged 65-80) with obesity and cardiometabolic risk factors .

DETAILED DESCRIPTION:
There is substantial evidence that overweight and obesity during late life (≥ 65 years of age) confers significant risk for type 2 diabetes and co-morbid conditions. Thus, there is growing concern about the public health consequences of increased incidence of type 2 diabetes in an aging United States population. Studies with high risk samples have shown that lifestyle interventions significantly reduce diabetes risk and that elders are particularly responsive, showing better weight loss and lower rates of diabetes development in comparison to younger individuals. However, although there have been program dissemination studies with mixed-age adult cohorts, few studies have focused specifically on persons ≥ 65 years of age or addressed the challenges of identifying workable platforms for delivering prevention programs to older adults. This application is based on the premise that offering an evidence-based lifestyle intervention to reduce risk for type 2 diabetes to retirees during the annual Medicare enrollment process presents an innovative, practical opportunity to reach eligible, high-risk adults. If shown to be feasible and effective, this program has strong potential for public health impact and medical cost-containment. Further, although clinical studies have emphasized the importance of continued contact over time in helping individuals extend the benefits of lifestyle interventions, there are no dissemination studies of which we are aware that have systematically documented the impact of continued monthly contacts after the initial intervention period. Thus, the overall aims of this application are to: 1. examine the feasibility and effectiveness of implementing the Group Lifestyle Balance 12-session program (GLB-12), an evidence-supported prevention program to mitigate diabetes risk, as part of the Medicare benefit offered to high risk retirees at a large public university, and; 2. evaluate the utility of continued telephone contact in enhancing treatment outcome at 12-months from baseline. Eligible participants will be 320 adults without diabetes, aged 65-80, with a BMI ≥ 27 and at least one additional cardiometabolic risk factor. All participants will receive the GLB-12 and then will be randomized to one of two continued contact protocols for the remaining one year of intervention, 8-sessions of continued small group contact by telephone (GLB-12 plus 8TC) or a newsletter control condition (GLB-12 plus NC). Program feasibility will be assessed by reporting enrollment, adherence and session completion rates, and satisfaction ratings in this delivery context. Effectiveness of the GLB-12 will be documented by reporting mean percent weight loss and the proportion of participants meeting ≥ 5% weight loss, a commonly accepted benchmark in translation studies known to be associated with favorable cardiometabolic outcomes at month 4. It also is hypothesized that GLB-12 plus 8TC, when compared to GLB-12 plus NC will be associated with more favorable anthropometric (weight, waist), cardiometabolic (glucose, blood pressure, lipid), physical function (chair stand, balance, gait speed) and health related quality of life outcomes at months 12 and 24. Finally, exploratory analyses will document program costs and program impact on medical utilization.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 65-80, with a BMI ≥ 27 and at least one of the following additional risk factors will be included: 1) Large waist circumference (> 40 inches men, >35 inches women) 2) hypertension or taking hypertension medication; 3) elevated lipids or taking medication for lipids or triglycerides 4) pre-diabetes (fasting glucose ≥ 100 mg/dL and < 126 mg/DL OR 5) or a score of 15 on the American Diabetes Association (ADA) risk test.

All study participants must have access to a telephone (including appropriate assistive devices if there are hearing impairments) and be able to read at the 6th grade level.

Exclusion Criteria:

* Individuals who report that they have been diagnosed by their doctor with diabetes or that they are taking any medicines used to treat diabetes
* lack of physician clearance for exercise participation before the 4th session
* a weight loss of 4.5 kgs or more in the past six months (to rule out unintentional weight loss that may be an indicator of current or incipient physical illness)
* current use of weight loss medications
* unable to attend at least 75% of the GLB 12-session program or are unwilling to self-monitor food, activity and weight as prescribed will be excluded and encouraged to consider joining in subsequent years.

Excluded individuals are referred to other clinical resources as appropriate.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 322 (Actual)
Dates: Start 2013-01-28 (Actual); Primary Completion 2017-05-26 (Actual); Study Completion 2017-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Venditti, PhD, Principal Investigator — University of Pittsburgh

IPD SHARING:
Plan to Share IPD: Yes
At the time of this R18 application in 2011 and resubmission and funding in 2012, a formal data sharing plan was neither required nor proposed. However, I will share final IPD with interested colleagues (including post-doctoral students and junior faculty, co-investigators at my institution across several departments including Medicine, Psychiatry, Epidemiology/Public Health). All data is de-identified per the original Data Safety and Monitoring Plan. All safeguards will be taken to ensure confidentiality and privacy of participants. I will not place limits on questions or methods of those sharing data files and only require that the Pitt Retiree Study participants and primary manuscripts resulting from this work, be acknowledged on all abstracts and manuscript publications resulting from the final data set.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The IPD, study protocol, informed consent form, and clinical study report will be available starting May 2019. No end date is specified.
Access Criteria: Contact the Principal Investigator directly at:
  vendittiem@upmc.edu

REFERENCES:
- [Background] Venditti EM, Marcus MD, Miller RG, Arena VC, Greenspan SL, Rockette-Wagner B. Group Lifestyle Phone Maintenance for Weight, Health, and Physical Function in Adults Aged 65-80 Years: A Randomized Clinical Trial. J Gerontol A Biol Sci Med Sci. 2021 Jan 18;76(2):352-360. doi: 10.1093/gerona/glaa229. PMID 32918078

RESULTS

PARTICIPANT FLOW:
Groups:
- GLB Plus Phone Contacts: GLB is the core behavioral lifestyle intervention delivered from 0-4 months using an in-person group format. The active comparator receives 8 additional sessions of group interactive telephone contact delivered from 5-12 months
  GLB plus phone contacts: GLB is a comprehensive evidence-based lifestyle intervention derived from the Diabetes Prevention Program intensive lifestyle intervention; combines behavior modification strategies and making health changes to diet, physical activity and weight. The active treatment group also receives 8 additional group phone conference calls for social support and problem solving.
- GLB Plus Newsletter Contacts: GLB is the core behavioral lifestyle intervention delivered from 0-4 months using in-person group format. The placebo comparator receives 4 additional educational newsletters delivered from 5-12 months.
  GLB plus newsletter contacts: GLB is a comprehensive evidence-based lifestyle intervention derived from the Diabetes Prevention Program intensive lifestyle intervention; combines behavior modification strategies and making health changes to diet, physical activity and weight. The placebo comparator includes 4 additional newsletters only.
Period: Overall Study
Arm/Group | GLB Plus Phone Contacts | GLB Plus Newsletter Contacts
Started | 162 | 160
Completed | 149 | 151
Not Completed | 13 | 9
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 13 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GLB Plus Phone Contacts | GLB Plus Newsletter Contacts | Total
Number analyzed (Participants) | 162 | 160 | 322
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (4.4) | 71.0 (4.2) | 71.2 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 121 | 247
  Male | 36 | 39 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 162 | 157 | 319
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 21 | 42
  White | 141 | 139 | 280
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms divided by meters squared] — Calculated as kilograms divided by meters squared
  kilograms divided by meters squared | 34.0 (5.6) | 33.5 (5.1) | 33.8 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Bodyweight
Description: Bodyweight of participant.
Time Frame: Change from baseline bodyweight at 12-months
Population: 162 participants were randomized to Group Lifestyle Balance (GLB) plus phone contacts and 160 were randomized to GLB plus newsletter contacts at 4 months. Of these 156 (96.3%) of GLB plus phone contacts and 156 (97.5%) of GLB plus newsletter contacts were included in the analysis of change in bodyweight at 12 months.
Measure: Mean (95% Confidence Interval); unit: percent weight change
Groups:
- Group Lifestyle Balance Plus Phone Contacts: Group Lifestyle Balance is the core behavioral lifestyle intervention delivered from 0-4 months using an in-person group format. The active comparator receives 8 additional sessions of group interactive telephone contact delivered from 5-12 months
  Group Lifestyle Balance plus phone contacts: Group Lifestyle Balance is a comprehensive evidence-based lifestyle intervention derived from the Diabetes Prevention Program intensive lifestyle intervention; combines behavior modification strategies and making health changes to diet, physical activity and weight. The active treatment group also receives 8 additional group phone conference calls for social support and problem solving.
- Group Lifestyle Balance Plus Newsletter Contacts: Group Lifestyle Balance is the core behavioral lifestyle intervention delivered from 0-4 months using in-person group format. The placebo comparator receives 4 additional educational newsletters delivered from 5-12 months.
  Group Lifestyle Balance plus newsletter contacts: Group Lifestyle Balance is a comprehensive evidence-based lifestyle intervention derived from the Diabetes Prevention Program intensive lifestyle intervention; combines behavior modification strategies and making health changes to diet, physical activity and weight. The placebo comparator includes 4 additional newsletters only.
Arm/Group | Group Lifestyle Balance Plus Phone Contacts | Group Lifestyle Balance Plus Newsletter Contacts
Number analyzed (Participants) | 156 | 156
percent weight change | -7.4 [-8.9 to -5.9] | -6.1 [-8.6 to -3.6]
Statistical Analysis 1: Comparison: Group Lifestyle Balance Plus Phone Contacts vs Group Lifestyle Balance Plus Newsletter Contacts; Test type: Superiority; p = 0.01, Mixed Models Analysis

2. Secondary Outcome: Change in Waist Circumference
Description: Waist circumference measured with a spring-loaded tape measure.
Time Frame: Change from baseline circumference at 12-months
Population: 162 participants were randomized to Group Lifestyle Balance (GLB) plus phone contacts and 160 were randomized to GLB plus newsletter contacts at 4 months. Of these 156 (96.3%) of GLB plus phone contacts and 156 (97.5%) of GLB plus newsletter contacts were included in the 12 month analysis of change in waist circumference.
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Group Lifestyle Balance Plus Phone Contacts | Group Lifestyle Balance Plus Newsletter Contacts
Number analyzed (Participants) | 156 | 156
cm | -5.3 [-6.4 to -4.2] | -4.1 [-6.8 to -1.4]
Statistical Analysis 1: Comparison: Group Lifestyle Balance Plus Phone Contacts vs Group Lifestyle Balance Plus Newsletter Contacts; Test type: Superiority; p = 0.15, Mixed Models Analysis

3. Secondary Outcome: Change in Fasting Total Cholesterol
Description: Total cholesterol (mg/dl) measured by finger-stick blood sample
Time Frame: Change from baseline level at 12-months
Population: 162 participants were randomized to Group Lifestyle Balance (GLB) plus phone contacts and 160 were randomized to GLB plus newsletter contacts at 4 months. Of these 156 (96.3%) of GLB plus phone contacts and 156 (97.5%) of GLB plus newsletter contacts were included in the analysis of change in fasting total cholesterol at 12 months.
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Group Lifestyle Balance Plus Phone Contacts | GLB Plus Newsletter Contacts
Number analyzed (Participants) | 156 | 156
mg/dl | -5.0 [-9.3 to -0.8] | -1.5 [-11.8 to 8.8]
Statistical Analysis 1: Comparison: Group Lifestyle Balance Plus Phone Contacts vs GLB Plus Newsletter Contacts; Test type: Superiority; p = 0.25, Mixed Models Analysis

4. Secondary Outcome: Change in Fasting High-Density Lipoprotein (HDL) Cholesterol
Description: HDL-cholesterol (mg/dl) measured by finger-stick blood sample
Time Frame: Change from baseline level at 12-months
Population: 162 participants were randomized to Group Lifestyle Balance (GLB) plus phone contacts and 160 were randomized to GLB plus newsletter contacts at 4 months. Of these, 156 (96.3%) GLB plus phone contacts and 156 (97.5%) GLB plus newsletter contacts were included in the analysis of change in fasting high-density lipoprotein cholesterol at 12 months.
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Group Lifestyle Balance Plus Phone Contacts | Group Lifestyle Balance Plus Newsletter Contacts
Number analyzed (Participants) | 156 | 156
mg/dl | 4.8 [3.2 to 6.4] | 2.9 [-1.1 to 6.9]
Statistical Analysis 1: Comparison: Group Lifestyle Balance Plus Phone Contacts vs Group Lifestyle Balance Plus Newsletter Contacts; Test type: Superiority; p = 0.11, Mixed Models Analysis

5. Secondary Outcome: Change in Fasting Low-Density Lipoprotein (LDL) Cholesterol
Description: LDL-cholesterol (mg/dl) measured by finger-stick blood sample
Time Frame: Change from baseline level at 12-months
Population: 162 participants were randomized to Group Lifestyle Balance (GLB) plus phone contacts and 160 were randomized to GLB plus newsletter contacts at 4 months. Of these 156 (96.3%) of GLB plus phone contacts and 156 (97.5%) of GLB plus newsletter contacts were included in the analysis of change in fasting Low-Density Lipoprotein (LDL) at 12 months.
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Group Lifestyle Balance Plus Phone Contacts | Group Lifestyle Balance Plus Newsletter Contacts
Number analyzed (Participants) | 156 | 156
mg/dl | -5.8 [-9.8 to -1.9] | -1.1 [-10.6 to 8.4]
Statistical Analysis 1: Comparison: Group Lifestyle Balance Plus Phone Contacts vs Group Lifestyle Balance Plus Newsletter Contacts; Test type: Superiority; p = 0.09, Mixed Models Analysis

6. Secondary Outcome: Change in Fasting Triglycerides
Description: Triglycerides (mg/dl) measured by fasting finger-stick sample
Time Frame: Change from baseline level at 12-months
Population: 162 participants were randomized to Group Lifestyle Balance (GLB) plus phone contacts and 160 were randomized to GLB plus newsletter contacts at 4 months. Of these 156 (96.3%) of GLB plus phone contacts and 156 (97.5%) of GLB plus newsletter contacts were included in the analysis of change in fasting triglycerides at 12 months.
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Group Lifestyle Balance Plus Phone Contacts | Group Lifestyle Balance Plus Newsletter Contacts
Number analyzed (Participants) | 156 | 156
mg/dl | -20.1 [-28.2 to -12.1] | -16.5 [-36.0 to 3.0]
Statistical Analysis 1: Comparison: Group Lifestyle Balance Plus Phone Contacts vs Group Lifestyle Balance Plus Newsletter Contacts; Test type: Superiority; p = 0.53, Mixed Models Analysis

7. Secondary Outcome: Change in Fasting Glucose
Description: Fasting glucose (mg/dl) measured by finger-stick sample
Time Frame: Change from baseline level at 12-months
Population: 162 participants were randomized to Group Lifestyle Balance (GLB) plus phone contacts and 160 were randomized to GLB plus newsletter contacts at 4 months. Of these 156 (96.3%) of GLB plus phone contacts and 156 (97.5%) of GLB plus newsletter contacts were included in the analysis of change in fasting glucose at 12 months.
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Group Lifestyle Balance Plus Phone Contacts | GLB Plus Newsletter Contacts
Number analyzed (Participants) | 156 | 156
mg/dl | -2.3 [-3.6 to -0.9] | -1.1 [-4.3 to 2.3]
Statistical Analysis 1: Comparison: Group Lifestyle Balance Plus Phone Contacts vs GLB Plus Newsletter Contacts; Test type: Superiority; p = 0.21, Mixed Models Analysis

8. Secondary Outcome: Change in Systolic Blood Pressure
Description: Systolic blood pressure (mmHg) measured by arm cuff digital blood pressure monitor (OMROM HEM90HXC)
Time Frame: Change from baseline level at 12-months
Population: 162 participants were randomized to Group Lifestyle Balance (GLB) plus phone contacts and 160 were randomized to GLB plus newsletter contacts at 4 months. Of these 156 (96.3%) of GLB plus phone contacts and 156 (97.5%) of GLB plus newsletter contacts were included in the analysis of change in systolic blood pressure at 12 months.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Group Lifestyle Balance Plus Phone Contacts | Group Lifestyle Balance Plus Newsletter Contacts
Number analyzed (Participants) | 156 | 156
mmHg | -2.6 [-5.2 to 0.004] | -1.6 [-8.0 to 4.7]
Statistical Analysis 1: Comparison: Group Lifestyle Balance Plus Phone Contacts vs Group Lifestyle Balance Plus Newsletter Contacts; Test type: Superiority; p = 0.60, Mixed Models Analysis

9. Secondary Outcome: Change in Diastolic Blood Pressure (mmHg)
Description: Diastolic blood pressure (mmHg) measured by arm cuff digital blood pressure monitor (OMROM HEM90HXC)
Time Frame: Change from baseline value at 12 months
Population: 162 participants were randomized to Group Lifestyle Balance (GLB) plus phone contacts and 160 were randomized to GLB plus newsletter contacts at 4 months. Of these 156 (96.3%) of GLB plus phone contacts and 156 (97.5%) of GLB plus newsletter contacts were included in the analysis of change in diastolic blood pressure at 12 months.
Measure: Mean (95% Confidence Interval); unit: mm/Hg
Arm/Group | Group Lifestyle Balance Plus Phone Contacts | Group Lifestyle Balance Plus Newsletter Contacts
Number analyzed (Participants) | 156 | 156
mm/Hg | -3.5 [-4.8 to -2.1] | -2.1 [-5.4 to 1.2]
Statistical Analysis 1: Comparison: Group Lifestyle Balance Plus Phone Contacts vs Group Lifestyle Balance Plus Newsletter Contacts; Test type: Superiority; p = 0.15, Mixed Models Analysis

10. Secondary Outcome: Change in Physical Function Performance Battery
Description: Short Physical Performance Battery (SPPB) total score (0-12) includes three function tests (each scored 0-4) and summed.
  The subtests are (1) gait speed measured in meters/second on a 4-meter walk route; (2) 3 progressive standing balance tests; (3) 5 chair stands. Higher score indicates better physical function.
Time Frame: Change from baseline score at 12-months
Population: 162 participants were randomized to Group Lifestyle Balance (GLB) plus phone contacts and 160 were randomized to GLB plus newsletter contacts at 4 months. Of these 156 (96.3%) of GLB plus phone contacts and 156 (97.5%) of GLB plus newsletter contacts were included in the analysis of change in the physical function performance battery at 12 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Lifestyle Balance Plus Phone Contacts | Group Lifestyle Balance Plus Newsletter Contacts
Number analyzed (Participants) | 156 | 156
score on a scale | 0.3 (1.4) | 0.3 (1.7)
Statistical Analysis 1: Comparison: Group Lifestyle Balance Plus Phone Contacts vs Group Lifestyle Balance Plus Newsletter Contacts; Test type: Superiority; p = 0.96, Mixed Models Analysis

11. Secondary Outcome: Change in Physical Activity Minutes/Week Using All CHAMPS Items
Description: Community Healthy Activities Model Program for Seniors (CHAMPS) physical activity questionnaire for older adults
Time Frame: Change from baseline minutes/week at 12-months
Population: 162 participants were randomized to Group Lifestyle Balance (GLB) plus phone contacts and 160 were randomized to GLB plus newsletter contacts at 4 months. Of these 155 (95.7%%) of GLB plus phone contacts and 156 (97.5%) of GLB plus newsletter contacts were included in the analysis of change in physical activity minutes /per week at 12 months.
Measure: Median (Inter-Quartile Range); unit: minutes/week
Arm/Group | Group Lifestyle Balance Plus Phone Contacts | Group Lifestyle Balance Plus Newsletter Contacts
Number analyzed (Participants) | 155 | 156
minutes/week | 30.0 [-165 to 300] | 30.0 [-225 to 323]
Statistical Analysis 1: Comparison: Group Lifestyle Balance Plus Phone Contacts vs Group Lifestyle Balance Plus Newsletter Contacts; Test type: Superiority; p = 0.96, Mixed Models Analysis

12. Secondary Outcome: Percentage Participants Achieving 3 or More Days of Moderate Intensity Physical Activities Per Week
Description: Stanford Brief Physical Activity categorical measure:
  Queries amount and intensity of typical weekly activities over the past month.
  1. most of week spent without any physical activity; sedentary at home; light chores; high intensity activities no more than 1-2 times per month.
  2. most days of week spent doing few activities; 1-2 times per week some light-moderate activity like walking or active chores at home.
  3. at least 3 times per week reports moderate activity such as brisk walking for 15-20 minutes or more, or at least 45-60 minutes of heavy home and yard chores.
  4. at least 3 times per week reports a regular program of moderate-vigorous intensity physical activities, or a regular program of fitness for 30 minutes or more, or active games like handball or tennis, or heavy home and yard chores for 60-minutes or more.
  Participants that endorse items 3 or 4 were considered to have achieved 3 or more days of moderate intensity physical activities per week.
Time Frame: percentage reporting higher intensity level activities 3 times per week or more at 12 months
Population: 162 participants were randomized to Group Lifestyle Balance (GLB) plus phone contacts and 160 were randomized to GLB plus newsletter contacts at 4 months. Of these, 155 (95.7%%) GLB plus phone contacts and 156 (97.5%) GLB plus newsletter contacts were included in analysis of percentage reporting higher intensity activities 3 times per week or more.
Measure: Count of Participants; unit: Participants
Arm/Group | Group Lifestyle Balance Plus Phone Contacts | Group Lifestyle Balance Plus Newsletter Contacts
Number analyzed (Participants) | 156 | 155
Participants | 110 | 81
Statistical Analysis 1: Comparison: Group Lifestyle Balance Plus Phone Contacts vs Group Lifestyle Balance Plus Newsletter Contacts; Test type: Superiority; p = 0.0009, Mantel Haenszel

13. Secondary Outcome: Change in Health Related Quality of Life-physical Component Summary Score
Description: Short-form 12-item health status questionnaire produces two scores: a physical component summary score and a mental component summary score. Scores range from 0-100 with higher scores indicating better health related quality of life. Each component score is transformed (standardized) using a mean of 50 and a standard deviation of 10.
Time Frame: Change from baseline score at 12-months
Population: 162 participants were randomized to Group Lifestyle Balance (GLB) plus phone contacts and 160 were randomized to GLB plus newsletter contacts at 4 months. Of these 156 (96.3%) of GLB plus phone contacts and 156 (97.5%) of GLB plus newsletter contacts were included in the analysis of change in health-related quality of life at 12 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Lifestyle Balance Plus Phone Contacts | Group Lifestyle Balance Plus Newsletter Contacts
Number analyzed (Participants) | 156 | 156
score on a scale | 2.26 (7.15) | 1.11 (7.74)
Statistical Analysis 1: Comparison: Group Lifestyle Balance Plus Phone Contacts vs Group Lifestyle Balance Plus Newsletter Contacts; Test type: Superiority; p = 0.18, Mixed Models Analysis

14. Secondary Outcome: Change in Nutrition
Description: Mediterranean Diet Assessment Tool. Total score ranges from 0 - 14. A higher score means higher adherence to a better quality of diet.
Time Frame: change from baseline score at 12-months
Population: 162 participants were randomized to Group Lifestyle Balance (GLB) plus phone contacts and 160 were randomized to GLB plus newsletter contacts at 4 months. Of these 156 (96.3%) of GLB plus phone contacts and 156 (97.5%) of GLB plus newsletter contacts were included in the analysis of change in Mediterranean Diet score at 12 months.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Group Lifestyle Balance Plus Phone Contacts | Group Lifestyle Balance Plus Newsletter Contacts
Number analyzed (Participants) | 156 | 156
score on a scale | 1 [0 to 2] | 1 [0 to 2]
Statistical Analysis 1: Comparison: Group Lifestyle Balance Plus Phone Contacts vs Group Lifestyle Balance Plus Newsletter Contacts; Test type: Superiority; p = 0.34, Mixed Models Analysis

15. Secondary Outcome: Change in Mood
Description: Center for Epidemiological Studies Depression Scale (CES-D) (score ranges 0-60; higher score indicates greater depressive symptoms)
Time Frame: change from baseline score at 12-months
Population: 162 participants were randomized to Group Lifestyle Balance (GLB) plus phone contacts and 160 were randomized to GLB plus newsletter contacts at 4 months. Of these 155 (95.7%) of GLB plus phone contacts and 155 (96.9%) of GLB plus newsletter contacts were included in the analysis of change in health-related quality of life at 12 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Lifestyle Balance Plus Phone Contacts | Group Lifestyle Balance Plus Newsletter Contacts
Number analyzed (Participants) | 155 | 155
score on a scale | 0.65 (5.44) | 0.49 (6.41)
Statistical Analysis 1: Comparison: Group Lifestyle Balance Plus Phone Contacts vs Group Lifestyle Balance Plus Newsletter Contacts; Test type: Superiority; p = 0.82, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse event data collected throughout the entire length of the study, 0 - 24 months.
Arm/Group | GLB Plus Phone Contacts | GLB Plus Newsletter Contacts
All-Cause Mortality (participants affected / at risk) | 0/162 | 1/160
Serious Adverse Events (participants affected / at risk) | 2/162 | 2/160
Other Adverse Events (participants affected / at risk) | 5/162 | 0/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLB Plus Phone Contacts (N=162) | GLB Plus Newsletter Contacts (N=160)
leg cellulitis (Infections and infestations) | 0 (0) | 1 (1)
inguinal hernia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
stroke (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLB Plus Phone Contacts (N=162) | GLB Plus Newsletter Contacts (N=160)
knee strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
gallstones (Gastrointestinal disorders) | 1 (1) | 0 (0)
aggravated spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
tendon tear from a fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study sample was predominantly white, female, middle-income and a single site study of urban and suburban communities in in southwestern Pennsylvania. Results may not generalize to other subgroups with high obesity-related health disparities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2012-05-24): https://cdn.clinicaltrials.gov/large-docs/75/NCT03192475/Prot_SAP_001.pdf
  • Informed Consent Form (2015-03-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT03192475/ICF_000.pdf